CLINICAL TRIAL: NCT01051479
Title: A Pilot C11-Choline PET-CT Imaging Study in Patients With Locally Advanced Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00012072; CCCWFU 60109 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Esophageal Cancer
Keywords: PET Positron emission tomography; CT X-ray computed tomography; Patients with Locally Advanced Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- C11-Choline (Experimental)
  Interventions: Drug: C11-Choline

INTERVENTIONS:
Drug: C11-Choline — 15 mCi 11C-choline will be administered intravenously as a bolus. The whole body emission scans will be acquired immediately following the tracer injection.

SUMMARY:
The purpose of this study is to evaluate the investigators ability to obtain reliable and meaningful 11C-Choline PET-CT images of esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or recurrent patients with locally advanced esophageal cancer with either squamous or adenocarcinoma histology.
* Ability to tolerate PET imaging
* Prior malignancy is allowed, but the expectation of survival must be that beyond that expected for patients with locally advanced esophageal cancer.

Exclusion Criteria:

* Pregnant or lactating females are not eligible for this pilot study.
* Patients having received chemotherapy in the 3 months prior to registration for any reason
* Patients with metastatic disease requiring chemoradiation for palliation are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To evaluate our ability to obtain reliable and meaningful 11C-Choline PET-CT images of esophageal cancer (pre- and post- chemotherapy). | 2 years

SECONDARY OUTCOMES:
Perform semi-quantitative analysis of tracer uptake using standard uptake values (SUV) and qualitative analysis using pure visual analysis. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States